CLINICAL TRIAL: NCT05718180
Title: Intrapartum Ultrasound for Assessment of Fetal Progression: a Randomised Controlled Trial to Evaluate the Variation of AoP, HSD, HPD, MLA, PAA According to Maternal Position and Pelvis (MaPP Study)
Brief Title: Intrapartum Ultrasound for Assessment of Fetal Progression
Acronym: Mapp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Mapp
Record Dates: First submitted 2022-05-06; First posted 2023-02-08 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Labor, Obstetric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine (Experimental): Measures are performed first in the supine position and then in a flexible sacrum position
  Interventions: Other: Transperineal imaging
- Flexible (Active Comparator): Measures are performed first in a kneeling squat position and then in the supine position
  Interventions: Other: Transperineal imaging

INTERVENTIONS:
Other: Transperineal imaging — To measure the difference between ultrasound parameters based on maternal position: to measure the variation of AoP (Angle of progression), MLA (Midline Angle), PAA(pubic arch angle expressed in grades) HSD (head-symphysis distance) HPD(head perineum distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the expulsion phase, in the resting step and during the push.

SUMMARY:
The use of ultrasound has been suggested to support the management of labour. According to several studies, ultrasound examination is more accurate and reproducible than clinical examination in diagnosing fetal head position, fetal station, and the prediction of labour arrest. Furthermore, there is growing evidence that ultrasound in labour may predict the outcome of instrumental vaginal delivery: a support to assess when an operative delivery is necessary. Ultrasound in labour can be performed using a transabdominal approach, mainly to determine head and spine position, or a transperineal approach, to assess head station and the situation at low stations. Several sonographic parameters have been proposed to evaluate the head station.

Furthermore, all ultrasound parameters studied so far, have always been measured with the woman in a supine position. While the biomechanics of childbirth with its mechanisms (known as nutation, counter-nutation of the pelvis, and the coccyx retropulsion) together with maternal movement, promote fetal rotation and the adaptation of its diameters with those of the maternal pelvis, allowing to gain more room for the fetal descent. Moreover, in most of the studies on intrapartum ultrasound, the mobility of the pelvis has not been mentioned. The contracted pelvis is the absence of mobility that leads to fetal-pelvic disproportion, arrest of labour, and operative delivery. Maternal pelvis biomechanics studies by high technological techniques have shown that maternal shifting positions during pregnancy and childbirth can create more room in the pelvis for safe delivery. The external and internal pelvic diameters are closely related.

For this reason, the evaluation of the mobility of the pelvis appears to be a necessary element to understand the ability of that pelvis to widen its diameters for fetal descent.

The aim of the study is to measure the variation of AoP, HSD, HPD, PAA in the supine position and in kneeling-squat position in the same woman and the cut-offs of the new ultrasound parameters and predictive capacity for vaginal birth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with singleton pregnancies
* at term gestation (37 weeks)
* fetus in cephalic presentation
* absence of factors hindering vaginal delivery

Exclusion Criteria:

* complicated pregnancies
* vaginal birth after Cesarean
* twin pregnancies
* early pregnancy
* women condition that exclude vaginal birth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound AoP EP | Beginning of the expulsive phase (active second stage): with complete dilation and the perception of an urge to push.
  To measure AoP (Angle of progression), expressed in degrees in the supine position and kneeling squat position in the same woman during the expulsion phase (EP) up to 3 hours
Ultrasound AoP RS | During the resting step
  To measure AoP (Angle of progression), expressed in degrees in the supine position and kneeling squat position in the same woman during the resting step (RS) up to 3 hours
Ultrasound AoP P | During the push
  To measure AoP (Angle of progression), expressed in degrees in the supine position and kneeling squat position in the same woman during the push (P) up to 3 hours
Ultrasound MLA EP | Beginning of the expulsive phase (active second stage): with complete dilation and the perception of an urge to push.
  To measure MLA (MidlineAngle) expressed in degrees in the supine position and kneeling squat position in the same woman during the expulsion up to 3 hours
Ultrasound MLA RS | During the resting step
  To measure MLA (MidlineAngle) expressed in degrees in the supine position and kneeling squat position in the same woman during the resting step up to 3 hours
Ultrasound MLA P | During the push
  To measure MLA (MidlineAngle) expressed in degrees in the supine position and kneeling squat position in the same woman during the push up to 3 hours
Ultrasound PAA EP | Beginning of the expulsive phase (active second stage): with complete dilation and the perception of an urge to push.
  To measure the PAA (pubic arch angle) expressed in degrees in the supine position and kneeling squat position in the same woman during the expulsion phase up to 3 hours
Ultrasound PAA RS | During the resting step
  To measure the PAA (pubic arch angle) expressed in degrees in the supine position and kneeling squat position in the same woman during the resting step up to 3 hours
Ultrasound PAA P | During the push
  To measure the PAA (pubic arch angle) expressed in degrees in the supine position and kneeling squat position in the same woman during the push up to 3 hours
Ultrasound HSD EP | Beginning of the expulsive phase (active second stage): with complete dilation and the perception of an urge to push.
  To measure the HSD (head-symphysis distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the expulsion phase up to 3 hours
Ultrasound HSD RS | During the resting step
  To measure the HSD (head-symphysis distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the resting step up to 3 hours
Ultrasound HSD P | During the push
  To measure the HSD (head-symphysis distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the push up to 3 hours
Ultrasound HPD EP | Beginning of the expulsive phase (active second stage): with complete dilation and the perception of an urge to push.
  To measure the HPD (head perineum distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the expulsion phase up to 3 hours
Ultrasound HPD RS | During the resting step
  To measure the HPD (head perineum distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the resting step up to 3 hours
Ultrasound HPD P | During the push
  To measure the HPD (head perineum distance) expressed in millimeters, in the supine position and kneeling squat position in the same woman during the push up to 3 hours

SECONDARY OUTCOMES:
mode of delivery | during delivery
  mode of delivery
duration of labour stages | during labour stages
  duration of labour stages up to 18 hours
fetal weight | at delivery
  fetal weight
fetal position | at the beginning of delivery
  fetal position
reasons for possible caesarean section | immediately after caesarean section
  reasons for possible caesarean section
Apgar Index at 1 min after delivery | One minute after delivery
  Apgar Index
Apgar Index 5 minutes after delivery | Five minutes after delivery
  Apgar Index
pH | Within 1 hour after delivery
  pH
BE | Within 1 hour after delivery
  Bases excess

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Ospedaliero Universitaria Sant'Orsola Malpighi, Bologna
  - Azienda Ospedale Università Padova, Padua
  - Ospedale Cristo Re, Roma